CLINICAL TRIAL: NCT07290959
Title: Indoor Daylight Photodynamic Therapy for Actinic Keratosis of the Scalp: Intra-patient Comparison Study of 1 Hour Versus 2 Hours Exposure Time
Brief Title: Indoor Daylight Photodynamic Therapy is an Effective, First-line Treatment for AK, But Its Feasibility is Limited by the Time Required for the Illumination (2 Hours). Our Objective Was to Evaluate the Efficacy of Idl-PDT With an Illumination Time of 1 Hour Versus 2 Hours in the Treatment of Scalp AK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Salvatore Hospital of L'Aquila (Other)
Responsible Party: Principal Investigator, Maria Esposito, Prof., San Salvatore Hospital of L'Aquila
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C.Et.R.A. 47/2025
Record Dates: First submitted 2025-11-17; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Actinic Keratosis (AK)
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AK patients (Experimental)
  Interventions: Other: We conducted an intra-patient, comparative study of idl-PDT with two illumination durations, 1 hour vs. 2 hours, using methyl aminolevulinate and a white LED light for the treatment of scalp AK.

INTERVENTIONS:
Other: We conducted an intra-patient, comparative study of idl-PDT with two illumination durations, 1 hour vs. 2 hours, using methyl aminolevulinate and a white LED light for the treatment of scalp AK. — The skin area to be treated was prepared with a sterile gauze pad soaked in saline solution to remove scales and crusts and then a 1 mm thick layer of cream containing 160mg/g of MAL (Metvix®) was applied. After 30 minutes of application, according to clinical practice and approved protocol, exposure to the white polychromatic LED lamp (Dermaris®, Surgiris, Croix, France, 400-700nm, fixed distance 30 cm, irradiance 72.6 W/m2) was performed, for a duration of 1 hour on one half and 2 hours on the other half, according to randomization. The emission spectrum of the light source was measured with a SR 9910 spectroradiometer (Macam Photometrics Ltd, Livingston, UK). The light doses were 26.1 J/cm2 for 1 hour illumination and 52.3 J/cm2 159 for 2 hours illumination, and the effective light doses for PpIX photoactivation were 0.69 Jeff/cm2 for 1 hour illumination and 1.39 Jeff/cm2 for 2 hours illumination. The effective light dose was calculated with the normalized PpIX absorption spectrum.

SUMMARY:
Several treatments are available for actinic keratosis (AK), many of which are hampered by local inflammation, pain, long duration, and slow healing. Indoor daylight photodynamic therapy (idl-PDT) is an effective, well-tolerated, first-line treatment for both AK and field cancerization, but the feasibility of this treatment is limited by the long time required for the illumination (2 hours). Objective of this study was to evaluate the efficacy of idl-PDT with an illumination time of 1 hour versus 2 hours in the treatment of scalp AK. Adult patients (age >50 years) with multiple AK located on the scalp (at least 5 Olsen grade I or II AK in two symmetrical areas) and diagnosed according to the typical clinical appearance were enrolled at two Dermatology Units in Italy. Exclusion criteria were the followings: previous treatment for AK within 6 months; status of congenital, infectious, or iatrogenic immunodepression; known cutaneous photosensitivity; known hypersensitivity to any ingredient of Metvix® 135 mg/g cream (Galderma SA, Lausanne, Switzerland). AK lesions on the scalp were mapped photographically with the support of a transparent sheet and graded according to Olsen grading scale. Two contralateral and symmetric areas of the scalp containing at least 5 AK were identified. Randomization of the two target areas for the two illumination durations (1 hour vs 2 hours) was performed with a 1:1 allocation ratio with a computer-generated list using permuted random blocks of six to ensure allocation concealment. At baseline, the following data were recorded: age, sex, phototype, Olsen grade and number of AK per side, any previous therapies on the treated area, any previous surgical excision of malignant skin neoplasms on the treated area, and comorbidities. The skin area to be treated was prepared with a sterile gauze pad soaked in saline solution to remove scales and crusts and then a 1 mm thick layer of cream containing 160mg/g of MAL (Metvix®) was applied. After 30 minutes of application, according to clinical practice and approved protocol, exposure to the white polychromatic LED lamp (Dermaris®, Surgiris, Croix, France, 400-700nm, fixed distance 30 cm, irradiance 72.6 W/m2 156 ) was performed, for a duration of 1 hour on one half and 2 hours on the other half, according to randomization. The emission spectrum of the light source was measured with a SR 9910 spectroradiometer (Macam Photometrics Ltd, Livingston, UK). The light doses were 26.1 J/cm2 for 1 hour illumination and 52.3 J/cm2 for 2 hours illumination, and the effective light doses for PpIX photoactivation were 0.69 Jeff/cm2 160 for 1 hour illumination and 1.39 Jeff/cm2 for 2 hours illumination. The effective light dose was calculated with the normalized PpIX absorption spectrum, the spectral irradiance of the lamps and treatment duration. Patients were evaluated 3 months and 6 months after the idl-PDT session to assess the efficacy of the two illumination times. A clinical photograph of the treated area was taken after 1 hour, 24 hours, and at each of the two follow-up visits. The primary endpoint of the study was the lesion response rate at 3 months. The analysis was performed on the total number of AK and after categorization of AK according to Olsen clinical grade. The secondary endpoints were lesion response rate at 6 months, tolerability and physicians' and patients' satisfaction. Tolerability was assessed as follows: subject's assessment of maximal pain perceived according to treated side immediately after the end of the treatment on a 0-10 numeric rating scale (NRS), from 0 (no pain) to 10 (extreme pain); local skin reactions (LSRs) assessed 1 hour and 24 hours after the treatment, including erythema, scaling, crusting, edema, blistering/pustulation and erosion/ulceration, each classified according to a 0-4 scale of severity (total LSR score range: 0-24). At the 3-months follow up visit, physicians rated their level of satisfaction on a 4-point scale with respect to treatment efficacy (very effective, effective, poorly effective, ineffective) and cosmetic outcome (excellent, good, poor or worse) for each treated area. In addition, patients were administered a questionnaire to globally assess convenience of the treatment (very convenient, convenient, poorly convenient, inconvenient) and overall level of satisfaction (very satisfied, satisfied, poorly satisfied, not satisfied at all) on a 4-point scale. The patient's willingness to undergo any further treatment with idl-PDT was recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >50 years) with multiple AK located on the scalp (at least 5 Olsen grade I or II AK in two symmetrical areas) and diagnosed according to their typical clinical dermoscopic appearance
* Subject must be able to understand and be willing to adhere to all protocol requirements and voluntarily sign and date an informed consent

Exclusion Criteria:

* previous treatment for AK within 6 months;
* status of congenital, infectious, or iatrogenic immunodepression;
* known cutaneous photosensitivity;
* known hypersensitivity to any ingredient of Metvix® 160 135 mg/g cream (Galderma SA, Lausanne, Switzerland).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study was the clinical clearance rate of actinic keratosis 3 months after the idl-PDT treatment, both overall and stratified by Olsen clinical grade | 3 months
  Treatment efficacy was measured by calculating the rate of complete clinical remission of actinic keratosis per 100 lesions-patient (defined by the number of completely responding actinic keratosis divided by the number of lesions treated at baseline) within each treated half. Comparison of treatment efficacy in the two halves (1h-half vs 2h-half) was analyzed by paired T-test. Statistical analysis was conducted with SPSS software (IBM) version 25.0 (SPSS Inc., Chicago, IL, USA). Differences were considered significant for p-values < 0.05.

SECONDARY OUTCOMES:
Pain perceived during the treatment, assessed with Numeric Pain Rating Scale (0-10) | Immediately after the end of the treatment
  The maximum pain perceived by the patients on each treated half was assessed using the Numerical Rating Scale (NRS) for pain, ranging from 0 (no pain) to 10 (extreme pain).
Cutaneous adverse events assessed with Local Skin Reactions (LSR) scale | 1 hour and 24 hours after the treatment
  Local skin reactions (LSRs) were assessed using LSR rating scale, considering six items (erythema, scaling, crusting, edema, blistering/pustulation and erosion/ulceration), each classified according to a 0-4 scale of severity (total LSR score range: 0-24).
Physicians' satisfaction to treatment efficacy | 3 months after the treatment
  Physicians rated their level of satisfaction on a 4-point scale with respect to treatment efficacy (very effective, effective, poorly effective, ineffective) for each treated area.
Physicians' satisfaction with cosmetic outcome | 3 months after the treatment
  Physicians rated their level of satisfaction on a 4-point scale with respect to cosmetic outcome (excellent, good, poor or worse) for each treated area.
Patients' global opinion on the treatment | 3 months after the treatment
  Patients were administered a questionnaire to globally assess their global opinion on the convenience of the treatment on a 4-point scale (very convenient, convenient, poorly convenient, inconvenient).
Patients' overall level of satisfaction | 3 months after the treatment
  Patients were administered a questionnaire to globally assess their overall level of satisfaction on the treatment on a 4-point scale (very satisfied, satisfied, poorly satisfied, not satisfied at all).

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Salvatore, L’Aquila, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antonetti P, Arisi M, Pellegrini C, Artelli GL, Zola A, Bruni M, Romano C, Galli B, Esposito M, Calzavara-Pinton P, Fargnoli MC. Indoor Daylight Photodynamic Therapy for Actinic Keratosis of the Scalp: Intrapatient Comparison Study of 1 h versus 2 h Exposure Time. Dermatol Ther (Heidelb). 2025 Dec 30. doi: 10.1007/s13555-025-01567-z. Online ahead of print. PMID 41467928